CLINICAL TRIAL: NCT02319395
Title: Behavioural Addiction and Genetics in Parkinson's Disease
Acronym: BADGE-PD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P100133
Record Dates: First submitted 2014-09-29; First posted 2014-12-18 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease; Impulse Control Disorders
Keywords: Parkinson's Disease; Behaviour addiction; Dopamine agonist; Genetic.
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One blood sampling during the study. A small number (1 to 5) of markers type "tag SNPs" or "coding SNP" will be selected for each of the selected genes, for a total of 50 markers (representing 20 to 25 genes). Non-silent coding SNP, that may have a functional effect, will be included as a priority. Genotyping is carried out by the method of genotyping VeraCode Goldengate.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cases: Presence of ICD in PD patients (cases) is defined as a score ≥ 2 at 1 hyperdopaminegic item, or 2 scores ≥ 2 at 1 hyperdopaminergic item of the scale for assessment of behavior and mood in PD (ECMP).
  Interventions: Genetic: Blood Sampling and DNA collection
- controls: Absence of ICD in PD patients (controls) is defined as a score ≤ 1 at all hyperdopaminergic items of ECMP and no more than 2 items of a score = 1.
  Interventions: Genetic: Blood Sampling and DNA collection

INTERVENTIONS:
Genetic: Blood Sampling and DNA collection — One blood sampling during the study. A small number (1 to 5) of markers type "tag SNPs" or "coding SNP" " (single nucleotide polymorphism, SNP) will be selected for each of the selected genes, for a total of 50 markers (representing 20 to 25 genes). Non-silent coding SNP, that may have a functional effect, will be included as a priority. Genotyping is carried out by the method of genotyping VeraCode Goldengate.

SUMMARY:
The " Behavioural Addiction and Genetics in Parkinson's Disease " study (BADGE-PD) is a national (France), multicenter, genetic association, case-control study to identify genetic factors associated with behavioural addiction (or Impulse Control Disorders, ICD) related to dopamine agonists treatment in Parkinson's disease (PD). Polymorphisms of candidate genes supposed to be involved in this adverse effect will be compared in 200 PD patients with ICD (n=200) and 200 matched PD patients without ICD (n=200).

DETAILED DESCRIPTION:
Objective: To identify susceptibility genes to impulse control disorders in Parkinson's Disease.

Study design: Genetic association study.

Primary objective:

To identify the susceptibility genes in behavior addiction in Parkinson's Disease

Secondary endpoints:

* To compare the clinical, neurological and psychiatric features of parkinsonian patients with behavior addiction compared to the control population. In case of differences between these groups, interaction will be studied with genetic factors
* Identify a psychometric profile from the TCI-R scale corresponding to the "hyperdopaminergic" subjects with AC personality

Patient selection:

Cases: patients with Parkinson's disease (PD) and impulse control disorder (ICD) as defined by a score greater than or equal to 2 or 3 scores greater than or equal to 2 at the "Evaluation Comportementale de la Maladie de Parkinson" scale (ECMP, Ardouin et al. 2009) for hyperdopaminergic items.

Controls: PD patients without impulse control disorder (ICD) as defined by a score of 0 or 1 at each hyperdopaminergic items AND no more than 2 items with a score of 1. Controls must have been treated with at least 300 mg of Levodopa equivalent daily dose for more than 12 months. Controls will be matched for sex, age, and age at onset of PD.

Number of subjects: 200 cases and 200 controls.

Clinical assessment: motor score (UPDRS), neuropsychological assessment, diagnostic criteria for addiction and ICD (MINI), self-administered psychometric questionnaire (TCI-R), treatment history, ICD history.

Genetic analysis: A blood sample will be taken for extraction and storage of DNA (DNA bank and Pitie-Salpetriere cells). Candidate genes* and polymorphisms will be selected from the literature data (receptors, transporters and metabolizing enzymes monoamine) and the molecular signature induced by L-DOPA in the striatum of a mice model of PD.

Statistical analysis:

A two-step analysis will be performed. For the first step, a training set (36% of subjects) will be analyzed with a logistic regression model considering an additive genetic effect. For the second step, the top 27% of the more significant genetic markers will be analyzed by using the left over replication set (64% of patients). Finally, a pooled analysis will be performed.

Sample Size: 200 patients per group to study 50 candidate markers with a power of 83% for genotype effect of 2.0, an additive genetic model, each allele frequency of 0.5.

* candidate genes list:

20 genes from the literature : DRD1, ANKK1, DRD2, DRD3, DRD4, DAT1, MAOA, COMT, HTR2A, HTR1B, TPH1, TPH2, 5HTT, GRIN2B, DBH, SCL6A2, BDNF, OPMR1, OPRK1, PDYN 8 genes from the experimentation: FosB, Arc, Nptx2, Ccrn4l, Car12, C8b, Mocs1, Mef2c

ELIGIBILITY:
Inclusion criteria :

Case Group

1. Age upper or equal to 30 years
2. Caucasian European (2 parents and 4 grandparents born in Europe)
3. Parkinson's disease according to the criteria of UKPDSBB
4. With a behavioral addiction defined as:

   * A score greater than or equal to 2 or 3 scores greater than or equal to 2 at hyperdopaminergic following items of Ardouin's scale (ECMP): eating behaviors, creativity, hobbyism, risk-taking behaviors, compulsive shopping, pathological gambling, hypersexuality, cyber-addiction, and Punding.
   * Onset under dopamine agonist or under L-DOPA
   * Present at the inclusion visit
   * OR in the past (<6 years). For these patients, the scale of Ardouin must have been passed at the time of behavior trouble or within 3 months after its disappearance.
5. Affiliation to a social security
6. Signature of the consent form

Control Group

1. Age upper or equal to 30 years
2. Caucasian European (2 parents and 4 grandparents born in Europe)
3. Parkinson's disease according to the criteria of UKPDSBB
4. Time evolution of the disease than or equal to 5 years
5. Having taken during its evolution a dopamine agonist dose at least equivalent to 300 mg of L-DOPA for at least 12 months.
6. Not having behavioral addiction

   * Not current, defined as a score of 0 or 1 and at most two items with a score of 1 on all items above and addiction to L-DOPA.
   * Neither passed, given authenticated by the semi-structured interview retrospective finding a score of 0 or 1 on all items hyperdopaminergic of Ardouin's scale (see above) AND no more than two items with a score of 1 and addiction to L-DOPA.
7. Affiliation to a social security
8. Signature of the consent form

Exclusion criteria :

Case Group

1. No Parkinson's disease or atypical parkinsonian syndrome
2. Taking neuroleptic except clozapine for patients with AC
3. Behavioral Addiction having started BEFORE taking the antiparkinsonian treatment

Control Group

1. No Parkinson's disease or atypical parkinsonian syndrome
2. Taking neuroleptic included clozapine for control patients
3. Behavioral Addiction having started BEFORE taking the antiparkinsonian treatment
4. Patient with guardianship, deprived of his liberty by judicial decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Allele frequency of 50 genetic markers (polymorphisms) will be compared between cases and controls. | baseline

SECONDARY OUTCOMES:
number of patients with a diagnostic of ICD according to the MINI | baseline
Total UPDRS (Unified Parkinson's Disease Rating Scale) score | baseline
Total score of the MMSE (Mini Mental State Examination) | baseline
Sub scores at the temperament and Character Inventory (revised version, TCI-R) | baseline
Number of subject in each group with personal or familial history of addiction | baseline

CONTACTS AND LOCATIONS:
Overall Officials: jean-christophe Corvol, MD, PhD, Principal Investigator — Assitance-Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier La Pitié Salpêtrière, Paris, France